CLINICAL TRIAL: NCT04556682
Title: Intravascular Lithotripsy and Rotational Atherectomy in Treatment of Severely Calcified Coronary Lesions
Brief Title: IVL and RA in Treatment of Balloon-crossable Severely Calcified Coronary Lesions
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Aboelkasem Ali Mousa, Assistant lecturer, Assiut University
Other Study IDs: IVL and RA in calcificaion
Record Dates: First submitted 2020-09-11; First posted 2020-09-21 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Coronary Calcification
Keywords: IVL; RA
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent Rotational atherectomy (RA): The device contains rapidly rotating burr that is coated with microscopic diamond chips, which debulks the calcified plaque by grinding the calcified atheroma into small particles facilitating stent passage and expansion. Both transfemoral or transradial approach can be used. Regular PCI guidewire can be used to cross the often complex anatomy then switching to a rotablation dedicated guidewire over a microcatheter. Burr sizes vary from 1.25mm up to 1.75mm (in certain cases bigger calibers may also be used) aiming to achieve plaque modification .
  Interventions: Device: Rotational atherectomy
- Patients who underwent Intravascular lithotripsy (IVL): The Coronary IVL System consists of an IVL Balloon Catheter with 2 integrated emitters, a Lithotripsy Generator, and a Connector Cable. These emitters create sonic pressure waves that selectively fracture calcium and alter vessel compliance facilitating stent passage and expansion. It is available in 2.5- to 4.0-mm diameters and 12 mm in length, with an inflation pressure of 4 atm used for delivering the treatment. Every catheter can emit a maximum of 80 pulses at a rate of one pulse per second. The IVL balloon catheter is chosen based on the reference lumen of the vessel and after pre-dilatation of the lesion (preferably with a non-compliant balloon) 10-30 pulses are given, usually with interval deflation to allow distal perfusion. If the lesion exceeds the 12 mm balloon length, the balloon can be repositioned and the IVL repeated .
  Interventions: Device: Intravascular lithotripsy

INTERVENTIONS:
Device: Rotational atherectomy — Device used for severely calcified coronary lesion preparation before stent implantation.
  Groups: Patients who underwent Rotational atherectomy (RA)
Device: Intravascular lithotripsy — Device used for severely calcified coronary lesion preparation before stent implantation.
  Groups: Patients who underwent Intravascular lithotripsy (IVL)

SUMMARY:
This study to compare periprocedural safety, angiographic success as well as short and long term outcomes of intravascular lithotripsy and rotational atherectomy as a method of severely calcified coronary lesion preparation before DES implantation.

DETAILED DESCRIPTION:
Coronary artery calcification (CAC) occurs in over 90% of men and 67% of women older than 70 years old .

Severe coronary calcification may be present in about 20% of patients undergoing percutaneous coronary intervention (PCI) .

Coronary calcification may impair stent delivery and expansion and damage the polymer/drug coating, resulting in impaired drug delivery and predispose to restenosis and stent thrombosis.

Intravascular imaging as intravascular ultrasound (IVUS) and optical coherence tomography (OCT) are good tools to assess calcium burden, distribution and thickness. Among the two imaging techniques, OCT was found to be more accurate than IVUS in defining calcium burden, calcium area , thickness and calcium length.

Rotational atherectomy (RA) as a method of severely calcified lesions modification before Drug-Eluting-Stent (DES) implantation has shown good outcomes in recent studies. However, its efficacy is reduced in presence of deep calcification.

Recently, intravascular lithotripsy (IVL) has been introduced as a novel modality for severely calcified coronary lesion preparation with good preliminary outcomes .

Currently the two techniques are regularly being used in combination in order to achieve optimal results . Whether IVL is a method equally good (or superior) to rotablation in cases where anatomy does not exclude the use of either technique (for example balloon-crossable, heavily calcified lesions) has not yet been discussed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years undergoing PCI because of stable angina (uncontrolled symptoms on optimal medical treatment) or post stabilized acute coronary syndrome (ACS).
* Patients have severe calcification: defined either angiographically or by OCT (or IVUS) as calcium arch >180º in at least one cross section , calcium length >5mm, calcium thickness >0.5 mm (2, 6).
* Vessel diameter ≥2.5mm and ≤4.0mm .
* Heavily calcified lesion length less than 40mm.
* All patients must have been discussed in the heart team of the hospital and accepted for coronary intervention

Exclusion Criteria:

* Severe coronary calcification with lesion uncrossable from a balloon.
* PCIs in the setting of STEMI or NSTEMI with persistent complains.
* Patients in cardiogenic shock.
* Heart failure New York Heart Association (NYHA) class IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease who found to have severe coronary calcification during percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Strategy success | Up to one day
  less than 20% in-stent residual stenosis of the target lesion and no postprocedural complications as no-reflow, dissection or perforation.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | after one year
  composite of Death, stroke, myocardial infarction, stent thrombosis, target vessel revascularization, and hospitalization at long term follow up

CONTACTS AND LOCATIONS:
Overall Officials: Amr youssef, professor, Study Chair — Assiut University; Johan W Jukema, professor, Study Chair — Leiden University Medical Center; Iannis Karalis, Doctor, Study Director — Leiden University Medical Center; Mohamed Abdelghany, professor, Study Chair — Assiut University; Salma M Taha, Lecturer, Study Chair — Assiut University; Mohamed AA Mousa, Doctor, Principal Investigator — Assiut University
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu W, Zhang Y, Yu CM, Ji QW, Cai M, Zhao YX, Zhou YJ. Current understanding of coronary artery calcification. J Geriatr Cardiol. 2015 Nov;12(6):668-75. doi: 10.11909/j.issn.1671-5411.2015.06.012. PMID 26788045
- [Background] Kassimis G, Didagelos M, De Maria GL, Kontogiannis N, Karamasis GV, Katsikis A, Sularz A, Karvounis H, Kanonidis I, Krokidis M, Ziakas A, Banning AP. Shockwave Intravascular Lithotripsy for the Treatment of Severe Vascular Calcification. Angiology. 2020 Sep;71(8):677-688. doi: 10.1177/0003319720932455. Epub 2020 Jun 22. PMID 32567327
- [Background] Bourantas CV, Zhang YJ, Garg S, Iqbal J, Valgimigli M, Windecker S, Mohr FW, Silber S, Vries Td, Onuma Y, Garcia-Garcia HM, Morel MA, Serruys PW. Prognostic implications of coronary calcification in patients with obstructive coronary artery disease treated by percutaneous coronary intervention: a patient-level pooled analysis of 7 contemporary stent trials. Heart. 2014 Aug;100(15):1158-64. doi: 10.1136/heartjnl-2013-305180. Epub 2014 May 20. PMID 24846971
- [Background] De Maria GL, Scarsini R, Banning AP. Management of Calcific Coronary Artery Lesions: Is it Time to Change Our Interventional Therapeutic Approach? JACC Cardiovasc Interv. 2019 Aug 12;12(15):1465-1478. doi: 10.1016/j.jcin.2019.03.038. PMID 31395217
- [Background] Lee MS, Shah N. The Impact and Pathophysiologic Consequences of Coronary Artery Calcium Deposition in Percutaneous Coronary Interventions. J Invasive Cardiol. 2016 Apr;28(4):160-7. Epub 2015 Aug 25. PMID 26301561
- [Background] Barbato E, Carrie D, Dardas P, Fajadet J, Gaul G, Haude M, Khashaba A, Koch K, Meyer-Gessner M, Palazuelos J, Reczuch K, Ribichini FL, Sharma S, Sipotz J, Sjogren I, Suetsch G, Szabo G, Valdes-Chavarri M, Vaquerizo B, Wijns W, Windecker S, de Belder A, Valgimigli M, Byrne RA, Colombo A, Di Mario C, Latib A, Hamm C; European Association of Percutaneous Cardiovascular Interventions. European expert consensus on rotational atherectomy. EuroIntervention. 2015 May;11(1):30-6. doi: 10.4244/EIJV11I1A6. PMID 25982648
- [Background] Kassimis G, Raina T, Kontogiannis N, Patri G, Abramik J, Zaphiriou A, Banning AP. How Should We Treat Heavily Calcified Coronary Artery Disease in Contemporary Practice? From Atherectomy to Intravascular Lithotripsy. Cardiovasc Revasc Med. 2019 Dec;20(12):1172-1183. doi: 10.1016/j.carrev.2019.01.010. Epub 2019 Jan 10. PMID 30711477
- [Background] Aksoy A, Salazar C, Becher MU, Tiyerili V, Weber M, Jansen F, Sedaghat A, Zimmer S, Leick J, Grube E, Gonzalo N, Sinning JM, Escaned J, Nickenig G, Werner N. Intravascular Lithotripsy in Calcified Coronary Lesions: A Prospective, Observational, Multicenter Registry. Circ Cardiovasc Interv. 2019 Nov;12(11):e008154. doi: 10.1161/CIRCINTERVENTIONS.119.008154. Epub 2019 Nov 11. PMID 31707803
- [Background] Jurado-Roman A, Gonzalvez A, Galeote G, Jimenez-Valero S, Moreno R. RotaTripsy: Combination of Rotational Atherectomy and Intravascular Lithotripsy for the Treatment of Severely Calcified Lesions. JACC Cardiovasc Interv. 2019 Aug 12;12(15):e127-e129. doi: 10.1016/j.jcin.2019.03.036. Epub 2019 Jul 17. No abstract available. PMID 31326422